CLINICAL TRIAL: NCT05577169
Title: Incorporating Mind-body Skills With Diabetes Education in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Tamara S. Hannon, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15268
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; Adolescent Behavior
Keywords: Type 1 diabetes; Adolescents; Mind-body skills
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The intervention will have two arms - one group will receive diabetes education with the addition of mind-body skills, and the other group will receive only diabetes education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-body skills + diabetes education (Experimental): Participants randomly assigned to this arm will undergo 20-30 minutes discussing a predetermined diabetes topic followed by 20-30 minutes working on a mind-body skills component. This mind-body skills component will be a combination of deep breathing, self-reflection, and meditation techniques focused on self-awareness to calm the stress-response. Participants will be assigned "homework" designed to encourage practice of the learned skill.
  Interventions: Behavioral: Mind-body skills; Behavioral: Diabetes education
- Diabetes education alone (Active Comparator): Participants randomly assigned to this arm will similarly undergo 20-30 minutes discussing the same predetermined diabetes topic as the intervention group.
  Interventions: Behavioral: Diabetes education

INTERVENTIONS:
Behavioral: Mind-body skills — The purpose of mind-body medicine is to use conscious thoughts and actions to positively impact autonomic responses from the brain as well as coping mechanisms for life's stresses. Examples of mind-body skills include deep breathing exercises, meditation, drawing, guided imagery, journaling, affirmations, and biofeedback.
  Arms: Mind-body skills + diabetes education
Behavioral: Diabetes education — When children and adolescents are diagnosed with diabetes, education is typically focused on the parents; as our older adolescents prepare to transition to adult care with full responsibility of their health, the goal of short education sessions is to review the basics of T1D along with addressing each individual's needs and questions as they make this transition.

SUMMARY:
Adolescence presents a challenging time for type 1 diabetes management, and despite a multitude of studies aimed at increasing disease compliance in this age group, none have been deemed superior. The purpose of this study is to incorporate mindfulness skills in with diabetes education sessions for adolescents with type 1 diabetes and study if this translates to improved outcomes in glycemic control, patient satisfaction, and mental wellness.

DETAILED DESCRIPTION:
This is a pilot study to learn if adding mind-body skills to diabetes education is useful in helping adolescents manage their type 1 diabetes. Specifically, the investigators will be studying adolescents aged 15-17 years old with uncontrolled diabetes defined by an A1c >9.0% who have also had the diagnosis of diabetes for at least 12 months. This study combines the teaching of mind-body skills with short virtual diabetes education sessions, in order to address both the direct needs of good diabetes management and the indirect needs of coping with diabetes-related stress and other external factors. The investigators will have two arms of the study - one receiving diabetes education with the addition of mind-body skills, and the other arm receiving only diabetes education. Sessions will be conducted virtually with 20-30 minutes of diabetes education, followed by 20-30 minutes of mind-body skills teaching in the respective arm. The study will consist of 10-12 weekly group sessions, with pre- and post-study questionnaires to evaluate mental and physical health. Participants will continue to attend their regular diabetes clinic appointments every three months. At the end of the study, participants will also partake in a short interview to gather feedback about their experience. The goals of this study are to evaluate the effect of mind-body skills as well as pilot test the feasibility and acceptability of such a project.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-17 years
* Diagnosis of type 1 diabetes for at least 12 months
* Uncontrolled diabetes with A1c at least 9.0%
* Parent or guardian agrees for adolescent to participate

Exclusion Criteria:

* Diagnosed cognitive disabilities
* Other uncontrolled chronic diseases as assessed by PI
* Inability to attend visits due to individual schedules

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention in the study population. | 12 months
  Feasibility of recruitment, retention of participants, and intervention completion. This will be measured by considering study participation rate, time to recruit, attendance, study retention rate, study completion rate, participant burden, and data completeness.
Acceptability of intervention in the study population. | 12 months
  This will be measured by participant satisfaction surveys.

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c, %) | 12 months
  The change in HbA1c will be measured from baseline to 12 months.

OTHER OUTCOMES:
Patient Health Questionnaire for Adolescents (PHQ-A) | 12 months
  Measure of general health and wellbeing. The change in the PHQ-A will be measured from baseline to 12 months.
Screen for Childhood Anxiety Related Emotional Disorders (SCARED-5) questionnaire | 12 months
  The change in the SCARED-5 will be measured from baseline to 12 months.
Problem Areas in Diabetes - Teens (PAID-T) questionnaire | 12 months
  The change in the PAID-T will be measured from baseline to 12 months.
Peds QL Diabetes Module questionnaire | 12 months
  The change in the Peds QL Diabetes Module will be measured from baseline to 12 months.
Mindful Attention Awareness Scale (MAAS) questionnaire for adolescents | 12 months
  The change in the MAAS will be measured from baseline to 12 months.
Difficulties in Emotion Regulation Scale (DERS) questionnaire | 12 months
  The change in the DERS will be measured from baseline to 12 months.
Child and Adolescent Social Support Scale (CASSS) questionnaire | 12 months
  The change in the parent and friends subscales of the CASSS will be measured from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara S. Hannon, MD, Principal Investigator — Riley Hospital for Children at Indiana University Health
Locations (2):
- United States (2):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No